CLINICAL TRIAL: NCT00314691
Title: Development of New Prenatal Diagnostic Tests From Maternal Blood
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Leaving of the person responsible for the data collection
Sponsor: University Hospital, Strasbourg, France (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3612
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2007-07

CONDITIONS: Hereditary Diseases
Keywords: fetal DNA; prenatal diagnosis; maternal plasma; Diagnostic potential of cell-free fetal DNA circulating in maternal blood
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Blood Specimen Collection

INTERVENTIONS:
Genetic: Blood samples

SUMMARY:
After extraction of the cell-free DNA circulating in maternal plasma, we aim at developing new techniques for fetal DNA enrichment to perform fetal gender determination, and indirect diagnosis of inherited diseases like Cystic Fibrosis, Huntington Disease, Myotonic Dystrophy, B-Thalassaemia...

ELIGIBILITY:
Inclusion Criteria:

* Mother and father-to-be both older than 18 years old
* Mother and father-to-be affiliated to social security
* Mother and father-to-be have good understanding of the protocol
* Pregnancy of the mother-to-be attested

Exclusion Criteria:

* Mother and father-to-be are younger than 18 years old
* Mother and/or father-to be refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Study Completion 2006-09

PRIMARY OUTCOMES:
Feasibility of fetal gender and genotype determination out of maternal blood

CONTACTS AND LOCATIONS:
Overall Officials: Romain FAVRE, MD, Principal Investigator — SIHCUS-CMCO de Schiltigheim, Strasbourg, FRANCE
Locations (1):
- Sihcus-Cmco, Strasbourg, Schiltigheim, France